CLINICAL TRIAL: NCT06983522
Title: The Effect of Toilet Training Awareness Program Given to Mothers
Brief Title: Providing Toilet Training Awareness Program to Mothers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muş Alparslan University (Other)
Collaborators: Ataturk University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: MusAlparslanU-YHB-İC-01
Record Dates: First submitted 2025-05-07; First posted 2025-05-21 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Implementation of Toilet Training Using Brazelton's Child-centered Approach
Keywords: toilet training; child; Brazelton Child-Centered Approach; parents; attitude
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Intervention Model Description: The experimental group and the control group were given toilet training.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: In the study, mothers who did not know which group they were in were blinded. Data were collected by a nurse working at the ASM who did not know which group she was collecting data from (blinded). Therefore, the researcher was also blinded. Since the groups were coded with numbers one and two in the SPSS program, statistical blinding was also applied.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Toilet Training (Experimental): 3 weeks old training program; In the 1st Stage of the training; Education on the subject of motherhood, the concept of motherhood and the role of motherhood.
  In the 2nd Stage of the training;Education on parental attitudes, types of attitudes.
  In the 3rd Stage of the training; Education on the subject of toilet training, the age of starting the training, the duration of the training, the signs of the child's readiness for toilet training, Brazelton's child-focused approach and the factors affecting toilet training, the effects of parental attitudes on toilet training and the problems that may be encountered during toilet training.
  Afterwards, Personal Information Form, Toilet Training BTÖ, ARÖ, ETÖ, scales will be presented.
  Interventions: Device: Toilet training booklet
- control group (No Intervention): No intervention was applied to the control group.

INTERVENTIONS:
Device: Toilet training booklet — Education on the subject of motherhood, the concept of motherhood and the role of motherhood. Education on parental attitudes, types of attitudes. Education on education in school, the age of starting education, the duration of education, signs of readiness for child toilet training, Brazelton's child-focused approach and characteristics of toilet training, the effects of parents' attitudes on toilet training and education on problems that may be encountered during toilet training. It covers the topics.
  Arms: Toilet Training

SUMMARY:
Toilet training has an important place among the developmental stages. A healthy child's ability to go to the toilet on his/her own is acquired between the ages of 1-3. Those who implement, show and guide toilet training have great responsibilities in ensuring that the period is healthy. Problems experienced during the education period can cause some negative situations, behaviors and undesirable personality traits in the child. The research will be conducted as an RCT in Muş Province, Family Health Center No. 01, between May 2024 and December 2025 in order to examine the effect of the toilet training awareness program applied to the participants on their knowledge and attitudes. The universe of the research will consist of participants who have not started 12-18 months of toilet training between May 2024 and May 2025. The entire universe will be examined in the research without using the sampling method. If the expected number cannot be reached between the specified dates and the relevant ASM, the data collection date will be extended. In the study, the Toilet Training Knowledge and Attitude Scale, the Motherhood Role Scale and the Parental Attitude Scale will be used to investigate the relationship between them. Children aged 12-18 months will be determined from the relevant ASM records. Phone numbers will be taken from the records, participants will be called and informed about the research and their verbal consent will be obtained. Participants who want to participate will be given an appointment and asked to come to ASM. Data will be obtained in the form of face-to-face interviews and questions and answers. Ethical principles will be followed.

DETAILED DESCRIPTION:
The aim of the study is to find out the effect of the toilet training awareness program applied to the participants on the knowledge and attitudes of the participants. There are many toilet training methods applied to date. Among these, the Child-Centered Approach developed by Brazelton is the most preferred. The American Academy of Pediatrics and the Canadian Pediatric Association also recommend this method. It is preferred more due to the presence of behaviors such as waiting for the child to be ready to start toilet training, having them do exercises, using positive terms and rewarding them if they are successful. Among the other applied methods, the ''One-Day Toilet Training'' method developed by Azrin and Fox was created for children with mental disabilities. It is less preferred due to behaviors such as harsh attitudes and verbal reprimands towards the child. Other methods such as Assisted Toilet Training or Elimination method are less preferred due to cultural differences or the constant observation and power required by mothers.

When we look at national and international studies, the knowledge levels of the participants are usually measured and their attitudes are evaluated. No toilet training program was applied to the participants. Therefore, the study is a first.

In this study, as researchers, we plan to create awareness in participants with children between the ages of 1-3 by giving them a toilet training program using Brazelton's Child-Centered Approach. In the study, the Toilet Training Knowledge and Attitude Scale, the Motherhood Role Scale and the Parenting Attitude Scale will be used to investigate the relationship between them.

ELIGIBILITY:
Inclusion Criteria:

* Being 12-18 months old,
* Being healthy (No growth and development problems, chronic diseases or hearing problems),
* Not having started toilet training

Exclusion Criteria:

* Mothers want to quit working,
* The child is diagnosed with a chronic disease and
* The mother cannot attend training.

Ages: 12 Months to 18 Months | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Mothers of childbearing age between the ages of 19-45
Enrollment: 83 (Actual)
Dates: Start 2025-01-07 (Actual); Primary Completion 2025-06-23 (Actual); Study Completion 2025-06-24 (Actual)

PRIMARY OUTCOMES:
Parental Attitude Scale | 3 months
  In the scale developed by Demir and Şendil in 2007, the scale consists of 46 items and four sub-dimensions. The scale is designed with a 5-point rating and the scores obtained from each dimension are calculated separately to obtain a score for each dimension. A high score obtained from the sub-dimensions indicates that the individual has the characteristic evaluated by the relevant sub-dimension. Cronbach alpha reliability coefficients were found as .83 for the democratic dimension, .76 for the authoritarian dimension, .75 for the overprotective dimension and .74 for the permissive dimension. One of these options is marked for each item. "Always like this" receives 5 points; "Mostly like this" receives 4 points; "Sometimes like this" receives 3 points; "Rarely like this" receives 2 points and "Never like this" receives 1 point.

SECONDARY OUTCOMES:
Toilet Training Knowledge Attitude Scale | 3 months
  It was developed by Ciger and Güdücü Tüfekci in 2019. It was developed to assess mothers' knowledge and attitudes during toilet training. The scale consists of 29 Likert-type items rated between 1 and 5 and does not contain reverse items or scoring. The highest score that can be obtained from the scale items is 5 and the lowest score is 1. (5-Strongly Agree, 4-Agree, 3-Don't Know, 2-Disagree, 1-Strongly Disagree). A high score shows that mothers have positive knowledge and attitudes. A minimum of 29 and a maximum of 145 points can be obtained from the scale. The Cronbach's α coefficient of Toilet Training-BTÖ was found to be .916. As the scale score increases, mothers' knowledge and attitudes towards Toilet Training-BTÖ increase positively.
Maternal Role Scale | 3 months
  It was developed by Arpacı Kızıldağ and Yiğit in 2022. The scale consists of 26 items and three sub-dimensions. There are 8 items in the Mother's Role sub-dimension, 11 items in the Mother's Attitude sub-dimension, and 7 items in the Mother's Concern sub-dimension. The scale was designed as "5-point Likert (1st Likert: Strongly Disagree, 2nd Likert: Disagree, 3rd Likert: Neither agree nor disagree, 4th Likert: Agree, 5th Likert: Strongly Agree)". The scoring of each item on the scale is 1-2-3-4-5. Items 7,8,9,10,14,15,19,20,21,22,23,24,25 on the scale are reverse coded. The scoring of these items will be 5-4-3-2-1. The maximum score obtained from the scale is 130 and the minimum score is 26, and increasing scores indicate that the motherhood role has developed. The "Cronbach's Alpha coefficient" of the scale was found to be 0.793.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma GÜDÜCÜ TÜFEKCİ, Prof.Dr., Study Director — fatma.guducutufekci@atauni.edu.tr
Locations (1):
- Family health center no. 01, Muş, Provincial, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I don't want to share